CLINICAL TRIAL: NCT04636008
Title: The Safety and Efficacy of Sintilimab Combined With Hypofractionated Radiotherapy in MSI-H/dMMR Rectal Cancer: a Prospective, Single-arm, Multicenter, Phase Ib Study
Brief Title: Sintilimab Plus Hypofractionated Radiotherapy for MSI-H/dMMR Rectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other); Yunnan Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Chengdu Third People's Hospital (Unknown); The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Meng Qiu, Prof., West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201919
Record Dates: First submitted 2020-11-11; First posted 2020-11-19 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Anti-PD-1 Antibody; Radiotherapy; Rectal Cancer; MSI-H; Mmr Deficiency
MeSH Terms: conditions — Rectal Neoplasms; Turcot syndrome | interventions — sintilimab; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Sintilimab+Hypofractionated radiotherapy
  Interventions: Drug: Sintilimab; Radiation: Hypofractionated Radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab+Hypofractionated radiotherapy
Radiation: Hypofractionated Radiotherapy — Hypofractionated Radiotherapy

SUMMARY:
This prospective, single-arm study is conducted to investigate the safety and efficacy of Sintilimab combined with hypofractionated radiotherapy in patients with microsatellite instability-high (MSI-H)/ DNA mismatch repair-deficient (dMMR) non-metastatic rectal cancer.

DETAILED DESCRIPTION:
The patients meet the inclusion criteria. After signing the informed consent, they are given radiotherapy 5Gyx5 and sintilimab 200mg ivgtt D1, D15, D29. Radical surgery is performed 6-8 weeks after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed rectal adenocarcinoma;
2. With DNA mismatch repair-deficient (dMMR) or microsatellite instability-high (MSI-H) status, whether or not being Lynch syndrome;
3. Not received any anti-rectal cancer treatment previously; for patients with Lynch syndrome, not received any anti-tumor therapy about rectal cancer diagnosed this time;
4. No distant metastasis except for lateral lymph nodes on thoracic and abdominal enhanced computed tomography (CT) scans; the distance between tumor's lower edge and anus within 15cm; clinical T stage ≥T2 on high-resolution pelvic magnetic resonance imaging (MRI)；
5. Men and women ≥18 years of age;
6. Eastern Cooperative Oncology Group performance status score 0 or 1;
7. Adequate hematologic, hepatic, renal, thyroid and cardiac function: hemoglobin ≥90 g/L, neutrophils ≥1500/mm3, platelets ≥75,000/mm3; aspartate aminotransferase and alanine aminotransferase ≤3.0 × upper limit of normal (ULN), bilirubin ≤1.5 × ULN; creatinine ≤1.5 × ULN, creatinine clearance ≥50 mL/min; activated partial thromboplastin time, prothrombin time and international normalized ratio ≤1.5 × ULN; serum albumin ≥28 g/L；thyroid stimulating hormone and free thyroxine within ±10% of normal levels; no obvious abnormality in electrocardiogram;
8. Not received blood, blood products and hematopoietic growth factor (e.g. granulocyte colony-stimulating factor) within 2 weeks before inclusion;
9. Informed consent form signed;
10. Life expectancy of ≥3 months.

Exclusion Criteria:

1. Allergic disease history, severe hypersensitivity to drugs, antibody products or Sintilimab;
2. Other malignancy history with disease free survival <5 years, except for curative in situ cervical cancer, curative skin basal cell carcinoma and curative gastrointestinal cancer by endoscopic mucoresection;
3. Current or past history of autoimmune diseases, including but not limited to: interstitial lung disease, uveitis, enteritis，active hepatitis (HBV DNA≥103 copies/mL after regular antiviral therapy)，nephritis, hyperthyroidism and hypothyroidism;
4. Immunosuppressant or corticosteroid (systemic or local) use to suppress immune function within 2 weeks before inclusion;
5. Severe infection needing intravenous antibiotics, antifungal agents or antiviral drugs, et al;
6. Congenital or acquired immunodeficiency such as HIV infection; active Hepatitis B (HBV DNA≥103 copies/mL after regular antiviral therapy);
7. Having one of the following complications: massive gastrointestinal hemorrhage, gastrointestinal perforation or obstruction; symptomatic heart diseases including unstable angina, myocardial infarction and heart failure; uncontrollable diabetes mellitus or hypertension; uncontrollable diarrhea (interfering with daily activities although receiving adequate treatment);
8. Bleeding tendency or receiving thrombolytic or anticoagulant therapy;
9. Pregnant or breastfeeding female; male and female unwilling to take any contraceptive measures;
10. Psychiatric disorders that would interfere with cooperation with the requirements of the study;
11. Other conditions that investigators consider not suitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Adverse reaction | up to 10 weeks
  Adverse reaction after receiving treatment of Sintilimab combined with hypofractionated radiotherapy and perioperative complications

SECONDARY OUTCOMES:
Pathological response rate | 6-8 weeks after radiotherapy
  Pathological response rate after treatment
Complete resection rate | 6-8 weeks after radiotherapy
  Complete resection rate after treatment
Quality of life questionnaire | up to 10 weeks
  Quality of life during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meng Qiu, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Li X, Fang C, Wang X, Yu Y, Wang Z, Qiu M. Neoadjuvant treatment of sintilimab plus hypofractionated radiotherapy for MSI-H/dMMR rectal cancer: A prospective, multicenter, phase Ib study. Cancer Med. 2022 Dec;11(23):4405-4410. doi: 10.1002/cam4.4720. Epub 2022 Mar 29. PMID 35352512